CLINICAL TRIAL: NCT00005543
Title: Genetic Epidemiology of Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 962-98; R01HL060279 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Cardiovascular Diseases; Venous Thromboembolism
MeSH Terms: conditions — Cardiovascular Diseases; Venous Thromboembolism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To determine the genetic epidemiology, including genetic and environmental interactions of the multifactorial disease, venous thromboembolism (VTE).

DETAILED DESCRIPTION:
BACKGROUND:

Venous thromboembolism is a major national health problem, with at least 201,000 first lifetime cases per year in the United States. Over 50,000 of these patients die within seven days, and for 20 percent, death is rapid, with insufficient time for medical intervention. Recurrent VTE is frequent and also associated with death as well as chronic impairment due to the venous stasis syndrome. Thus, identification of high-risk patients for targeted VTE prophylaxis or treatment is necessary to improve survival and prevent impairment. While clinical risk factors can identify a population at risk, such risk factors have low predictive value for the individual patient. The high prevalence of the Factor V R506Q (Leiden) and Prothrombin 20210G --> A mutations among VTE patients suggests the hypothesis that additional genetic abnormalities of coagulation (thrombophilia) are associated with a substantial proportion of VTE cases.

DESIGN NARRATIVE:

The study had a case-control design. Using stored DNA samples, the investigators screened for mutations within the candidate genes for Factor V R506Q (Leiden) and Prothrombin 20210G --> A using either dideoxy, bi-directional dideoxy, or restriction endonuclease fingerprinting, and performing population-based case-control and cohort studies using a previously identified 30-year VTE inception cohort.

The specific aims were: 1) to screen genomic DNA from patients with VTE for mutations within (candidate) genes encoding for prothrombin, thrombomodulin, tissue factor pathway inhibitor, tissue factor, factor VII, and factor X, and to determine if the mutation predicted a change in either protein expression or structure; 2) in population-based case-control studies, a) to test the hypothesis that such a mutation was associated with VTE, estimate the strength of the association, and determine the independence of the association after controlling for other environmental risk factors and coagulation abnormalities, including interactions, and b) to test the hypothesis that a mutation was associated with death and autopsy; 3) to estimate the attributable risk for VTE associated with each significant mutation, both individually and for all independently significant mutations collectively while controlling for other environmental risk factors and coagulation abnormalities; and 4) in a population-based retrospective cohort study, to estimate the time-to-VTE recurrence and to test the hypothesis that each significant mutation was an independent predictor of VTE recurrence after controlling for other environmental predictors and coagulation abnormalities, including interactions.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3135 (Actual)
Dates: Start 1999-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Heit — Mayo Foundation

REFERENCES:
- [Background] Taliani MR, Roberts SC, Dukek BA, Pruthi RK, Nichols WL, Heit JA. Sensitivity and specificity of denaturing high-pressure liquid chromatography for unknown protein C gene mutations. Genet Test. 2001 Spring;5(1):39-44. doi: 10.1089/109065701750168680. PMID 11336399
- [Background] Heit JA. Prevention of venous thromboembolism. Clin Geriatr Med. 2001 Feb;17(1):71-92. doi: 10.1016/s0749-0690(05)70107-5. PMID 11270135
- [Background] Shields RC, McBane RD, Kuiper JD, Li H, Heit JA. Efficacy and safety of intravenous phytonadione (vitamin K1) in patients on long-term oral anticoagulant therapy. Mayo Clin Proc. 2001 Mar;76(3):260-6. doi: 10.4065/76.3.260. PMID 11243272
- [Background] Swensen SJ, Sheedy PF 2nd, Ryu JH, Pickett DD, Schleck CD, Ilstrup DM, Heit JA. Outcomes after withholding anticoagulation from patients with suspected acute pulmonary embolism and negative computed tomographic findings: a cohort study. Mayo Clin Proc. 2002 Feb;77(2):130-8. doi: 10.4065/77.2.130. PMID 11838646
- [Background] Heit JA. Perioperative management of the chronically anticoagulated patient. J Thromb Thrombolysis. 2001 Sep;12(1):81-7. doi: 10.1023/a:1012746729537. PMID 11711693
- [Background] Heit JA, Rooke TW, Silverstein MD, Mohr DN, Lohse CM, Petterson TM, O'Fallon WM, Melton LJ 3rd. Trends in the incidence of venous stasis syndrome and venous ulcer: a 25-year population-based study. J Vasc Surg. 2001 May;33(5):1022-7. doi: 10.1067/mva.2001.113308. PMID 11331844
- [Background] Heit JA. Low-molecular-weight heparin: the optimal duration of prophylaxis against postoperative venous thromboembolism after total hip or knee replacement. Thromb Res. 2001 Jan 1;101(1):V163-73. doi: 10.1016/s0049-3848(00)00388-1. PMID 11342096
- [Background] Danilenko-Dixon DR, Heit JA, Silverstein MD, Yawn BP, Petterson TM, Lohse CM, Melton LJ 3rd. Risk factors for deep vein thrombosis and pulmonary embolism during pregnancy or post partum: a population-based, case-control study. Am J Obstet Gynecol. 2001 Jan;184(2):104-10. doi: 10.1067/mob.2001.107919. PMID 11174488
- [Background] Heit JA. Venous thromboembolism epidemiology: implications for prevention and management. Semin Thromb Hemost. 2002 Jun;28 Suppl 2:3-13. doi: 10.1055/s-2002-32312. PMID 12073175
- [Background] Heit JA. Mapping out the future in venous thromboembolism and acute coronary syndromes. Semin Thromb Hemost. 2002 Aug;28 Suppl 3:33-9. doi: 10.1055/s-2002-34073. PMID 12232821
- [Background] Heit JA. Risk factors for venous thromboembolism. Clin Chest Med. 2003 Mar;24(1):1-12. doi: 10.1016/s0272-5231(02)00077-1. PMID 12685052
- [Background] Heit JA. Current management of acute symptomatic deep vein thrombosis. Am J Cardiovasc Drugs. 2001;1(1):45-50. doi: 10.2165/00129784-200101010-00005. PMID 14728051
- [Background] Heit JA, Petterson TM, Owen WG, Burke JP, DE Andrade M, Melton LJ 3rd. Thrombomodulin gene polymorphisms or haplotypes as potential risk factors for venous thromboembolism: a population-based case-control study. J Thromb Haemost. 2005 Apr;3(4):710-7. doi: 10.1111/j.1538-7836.2005.01187.x. PMID 15842356
- [Background] Heit JA, Sobell JL, Li H, Sommer SS. The incidence of venous thromboembolism among Factor V Leiden carriers: a community-based cohort study. J Thromb Haemost. 2005 Feb;3(2):305-11. doi: 10.1111/j.1538-7836.2004.01117.x. PMID 15670037